CLINICAL TRIAL: NCT04088474
Title: Functional Assessment in The Intestinal Flora Improvement
Brief Title: Effects of Vigiis 101-LAB on a Healthy Populations' Gut Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Sunway002
Record Dates: First submitted 2019-09-05; First posted 2019-09-12 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Microbiome
Keywords: gut microflora; Lactobacillus paracasei subsp. paracasei NTU 101; probiotics

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, placebo-controlled clinical study
Who Masked: Participant
Masking Description: a randomized, double-blind, placebo-controlled clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vigiis 101-LAB (Experimental): The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were made into capsules (Vigiis 101-LAB capsule I) containing 5 billion bacteria per capsule for the gut flora clinical trial. The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were also mixed into capsules (Vigiis 101- LAB capsule II) containing 5 billion bacteria per capsule for clinical trial.
  Interventions: Dietary Supplement: Vigiis 101-LAB
- placebo (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vigiis 101-LAB — examined the effects of the Vigiis 101-LAB capsules (5 billion CFU/day)
  Arms: Vigiis 101-LAB
Dietary Supplement: Placebo — Maltodextrin was used as a placebo
  Arms: placebo

SUMMARY:
This clinical trial was conducted as part of the "Methods for Evaluating the Improvement of Gastrointestinal Function in Health Food" announced by the Department of Health, DOH (currently known as Ministry of Health and Welfare, MOHW) on the test article, "Vigiis 101-LAB powder (Capsules)", manufactured by SunWay Biotech Co., Ltd.

DETAILED DESCRIPTION:
1.1 Introduction The human microbiome comprises diverse microbiologic ecosystems and is composed of a variety of bacteria, archaea, microeukaryotes, and viruses. Although investigators have appreciated the diversity of our microbial world for decades, scientists were constrained by the inability to culture many bacteria in the laboratory. Paradigms in biomedical science and medicine are changing in a fundamental way as investigators explore potential contributions of human-associated microbes to health and expand our understanding of disease susceptibility and pathogenesis. In the 21st century, investigators are attempting to develop a more balanced mindset as investigators seek to understand the role of the human microbiome in physiology and manipulate it to optimize health and prevent or treat disease. In recent years, investigators have increased our understanding of microbial communities and their corresponding metagenomes at different human body sites greatly. Healthy gastrointestinal (GI) microbiome should include age, sex, race/ethnicity, and diet. The Human Microbiome Project documented the importance of considering sex and race/ethnicity in evaluating differences between microbiomes of individuals. The human GI microbiome comprises diverse microbial communities that differ based on their location along the length of the GI tract (esophagus, stomach, small intestine, and large intestine or colon). Most human intestinal microbiome studies have relied on stool specimens. Probiotics have showed to possess anti mutagenic, anti carcinogenic and hypocholesterolemic properties. It is well-known that probiotics have a number of beneficial health effects in humans and animals, including the reduction of symptoms in lactose intolerance and enhancement of the bio availability of nutrients. Further, they were also observed to have antagonistic actions against intestinal and food-borne pathogens, to decrease the prevalence of allergies in susceptible individuals and to have immunomodulatory effects. Typically, the bacteria colonise the intestinal tract first and then reinforce the host defence systems by inducing a generalised mucosal immune response, balanced T-helper cell response, self-limited inflammatory response and secretion of polymeric IgA. Scientific reports showed that the Taiwan native lactic acid bacterium from newborn infant faeces identified as Lactobacillus paracasei subsp. paracasei NTU 101 and its fermented products proved to be effective for the management of blood cholesterol and pressure, prevention of gastric mucosal lesion development, immunomodulation and alleviation of allergies, anti-osteoporosis and inhibition the fat tissue accumulation.

1.2 Materials The strain used in the current study was L. paracasei subsp. paracasei NTU 101 (lyophilized powdered, Vigiis 101-LAB; probiotic powder from SunWay Biotech Co., Ltd., Taipei, Taiwan). The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were made into capsules (Vigiis 101-LAB capsule) containing 5 billion bacteria per capsule for the gut flora clinical trial. Maltodextrin was used as a placebo.

1.3 Randomized, double-blind clinical criteria of effects of Vigiis 101-LAB capsule I on gut flora (clinical trial) Vigiis 101-LAB capsule was administered orally once per day, one capsule each time. The entire study took 4 weeks, and subjects were prohibited from eating fermented food products, such as miso, kimchi, fermented dairy products, oligosaccharide-containing foods, and lactic acid bacteria-containing products. Subjects also avoided consuming excessive gas-producing foods (such as soybeans and sweet potatoes) during their daily meals and avoided foods that can cause abdominal distension or promote peristalsis (such as lactic acid beverages and oligosaccharide-containing beverages). After the trial started, subjects recorded their daily number of bowel movements and completed relevant questionnaires at weeks 0, 2, and 4. The subjects visited the doctor once every 2 weeks for monitoring gastrointestinal function and physiological characteristics. At weeks 0, 1, 2, 3, and 4, fecal samples from the subjects were collected and put into bottles containing an anaerobic diluent and shaken to uniformly mix the feces and diluent.

1.4 Outcome measurements Fecal moisture content and pH value testing. Blood biochemical tests were carried out in the laboratory.

1.5. Statistical analysis Data are expressed as the mean ± standard deviation (SD). The statistical significance of the biochemical analyses was determined by one-way analysis of variance (ANOVA) using the general linear model procedure of the statistical product and service solutions software (SPSS Institute, Inc., Chicago, IL, USA). This was followed by ANOVA with a paired t-test to evaluate the difference before and after sample and placebo administration, while the Student t-test was used to compare the difference between test and placebo groups (P ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≧ 20 years and ≦ 65 years.
2. Subjects with normal weight (body mass index: 18.5-24).
3. Subjects with no gastrointestinal diseases or on medication.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects who are allergic to Lactobacillus.
3. Subjects with chronic gastrointestinal diseases.
4. Subjects who previously underwent gastrectomy or gastric bypass.
5. Subjects with liver, kidney, or heart disease, alcoholism, or uncontrolled diabetes.
6. Subjects who developed stroke, psychiatric diseases, or depression within the last 1 year.
7. Subjects being administered drugs that can regulate gastrointestinal function, functional foods, bacteriostatic drugs or supplements, antibiotics, antioxidants, or other unknown drugs within the last 2 weeks.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-12-18 (Actual)

PRIMARY OUTCOMES:
Microflora analysis of fecal contents | 4 week
  culture for intestinal defecation Bifidobacterium spp. Clostridium perfringens. Lactobacillus spp. and Escherichia coli

CONTACTS AND LOCATIONS:
Overall Officials: Jyh Ming Liou, MD,PHD, Study Director — National Taiwan University Hospital; Tsong Ming Lu, MD, Principal Investigator — Cheng Hsin Hospital
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine, National Taiwan University Hospital, National Taiwan University College of Medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Effects of Vigiis 101-LAB capsule on improving gut microflora was examined
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Medicine / Nursing Medical Doctor Healthcare / Medical Management Medical Technician Pharmacist Nurse / Nursing Personnel Clinical Coodinator Clinical Researcher

REFERENCES:
- [Result] Agace WW, McCoy KD. Regionalized Development and Maintenance of the Intestinal Adaptive Immune Landscape. Immunity. 2017 Apr 18;46(4):532-548. doi: 10.1016/j.immuni.2017.04.004. PMID 28423335
- [Result] Arnao MB, Cano A, Hernandez-Ruiz J, Garcia-Canovas F, Acosta M. Inhibition by L-ascorbic acid and other antioxidants of the 2.2'-azino-bis(3-ethylbenzthiazoline-6-sulfonic acid) oxidation catalyzed by peroxidase: a new approach for determining total antioxidant status of foods. Anal Biochem. 1996 May 1;236(2):255-61. doi: 10.1006/abio.1996.0164. PMID 8660502
- [Result] Atarashi K, Tanoue T, Shima T, Imaoka A, Kuwahara T, Momose Y, Cheng G, Yamasaki S, Saito T, Ohba Y, Taniguchi T, Takeda K, Hori S, Ivanov II, Umesaki Y, Itoh K, Honda K. Induction of colonic regulatory T cells by indigenous Clostridium species. Science. 2011 Jan 21;331(6015):337-41. doi: 10.1126/science.1198469. Epub 2010 Dec 23. PMID 21205640
- [Result] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Result] Belkaid Y, Harrison OJ. Homeostatic Immunity and the Microbiota. Immunity. 2017 Apr 18;46(4):562-576. doi: 10.1016/j.immuni.2017.04.008. PMID 28423337
- [Result] Bengmark S. Gut microbiota, immune development and function. Pharmacol Res. 2013 Mar;69(1):87-113. doi: 10.1016/j.phrs.2012.09.002. Epub 2012 Sep 16. PMID 22989504
- [Result] Bridgman SL, Azad MB, Field CJ, Haqq AM, Becker AB, Mandhane PJ, Subbarao P, Turvey SE, Sears MR, Scott JA, Wishart DS, Kozyrskyj AL; CHILD Study Investigators. Fecal Short-Chain Fatty Acid Variations by Breastfeeding Status in Infants at 4 Months: Differences in Relative versus Absolute Concentrations. Front Nutr. 2017 Apr 10;4:11. doi: 10.3389/fnut.2017.00011. eCollection 2017. PMID 28443284
- [Result] Chen T, Isomaki P, Rimpilainen M, Toivanen P. Human cytokine responses induced by gram-positive cell walls of normal intestinal microbiota. Clin Exp Immunol. 1999 Nov;118(2):261-7. doi: 10.1046/j.1365-2249.1999.01047.x. PMID 10540188
- [Result] Kopp-Hoolihan L. Prophylactic and therapeutic uses of probiotics: a review. J Am Diet Assoc. 2001 Feb;101(2):229-38; quiz 239-41. doi: 10.1016/S0002-8223(01)00060-8. PMID 11271697
- [Result] Krasowska A, Sigler K. How microorganisms use hydrophobicity and what does this mean for human needs? Front Cell Infect Microbiol. 2014 Aug 19;4:112. doi: 10.3389/fcimb.2014.00112. eCollection 2014. PMID 25191645
- [Result] Lee N, Kim WU. Microbiota in T-cell homeostasis and inflammatory diseases. Exp Mol Med. 2017 May 26;49(5):e340. doi: 10.1038/emm.2017.36. PMID 28546563
- [Result] Dement JM, Epling C, Joyner J, Cavanaugh K. Impacts of Workplace Health Promotion and Wellness Programs on Health Care Utilization and Costs: Results From an Academic Workplace. J Occup Environ Med. 2015 Nov;57(11):1159-69. doi: 10.1097/JOM.0000000000000555. PMID 26539763
- [Result] Lin FM, Chiu CH, Pan TM. Fermentation of a milk-soymilk and Lycium chinense Miller mixture using a new isolate of Lactobacillus paracasei subsp. paracasei NTU101 and Bifidobacterium longum. J Ind Microbiol Biotechnol. 2004 Dec;31(12):559-64. doi: 10.1007/s10295-004-0184-z. Epub 2004 Nov 18. PMID 15662546
- [Result] Liu CF, Tung YT, Wu CL, Lee BH, Hsu WH, Pan TM. Antihypertensive effects of Lactobacillus-fermented milk orally administered to spontaneously hypertensive rats. J Agric Food Chem. 2011 May 11;59(9):4537-43. doi: 10.1021/jf104985v. Epub 2011 Apr 4. PMID 21446645
- [Result] Lobo V, Patil A, Phatak A, Chandra N. Free radicals, antioxidants and functional foods: Impact on human health. Pharmacogn Rev. 2010 Jul;4(8):118-26. doi: 10.4103/0973-7847.70902. PMID 22228951
- [Result] Miller NJ, Sampson J, Candeias LP, Bramley PM, Rice-Evans CA. Antioxidant activities of carotenes and xanthophylls. FEBS Lett. 1996 Apr 22;384(3):240-2. doi: 10.1016/0014-5793(96)00323-7. PMID 8617362
- [Result] Naidu AS, Bidlack WR, Clemens RA. Probiotic spectra of lactic acid bacteria (LAB). Crit Rev Food Sci Nutr. 1999 Jan;39(1):13-126. doi: 10.1080/10408699991279187. PMID 10028126
- [Result] Orrhage K, Sillerstrom E, Gustafsson JA, Nord CE, Rafter J. Binding of mutagenic heterocyclic amines by intestinal and lactic acid bacteria. Mutat Res. 1994 Dec 1;311(2):239-48. doi: 10.1016/0027-5107(94)90182-1. PMID 7526189
- [Result] Ouwehand AC, Isolauri E, Kirjavainen PV, Tolkko S, Salminen SJ. The mucus binding of Bifidobacterium lactis Bb12 is enhanced in the presence of Lactobacillus GG and Lact. delbrueckii subsp. bulgaricus. Lett Appl Microbiol. 2000 Jan;30(1):10-3. doi: 10.1046/j.1472-765x.2000.00590.x. PMID 10728552
- [Result] Ouwehand AC, Salminen S, Isolauri E. Probiotics: an overview of beneficial effects. Antonie Van Leeuwenhoek. 2002 Aug;82(1-4):279-89. PMID 12369194
- [Result] Pant N, Marcotte H, Brussow H, Svensson L, Hammarstrom L. Effective prophylaxis against rotavirus diarrhea using a combination of Lactobacillus rhamnosus GG and antibodies. BMC Microbiol. 2007 Sep 27;7:86. doi: 10.1186/1471-2180-7-86. PMID 17900343
- [Result] Perdigon G, Vintini E, Alvarez S, Medina M, Medici M. Study of the possible mechanisms involved in the mucosal immune system activation by lactic acid bacteria. J Dairy Sci. 1999 Jun;82(6):1108-14. doi: 10.3168/jds.S0022-0302(99)75333-6. PMID 10386296
- [Result] Pool-Zobel BL, Neudecker C, Domizlaff I, Ji S, Schillinger U, Rumney C, Moretti M, Vilarini I, Scassellati-Sforzolini R, Rowland I. Lactobacillus- and bifidobacterium-mediated antigenotoxicity in the colon of rats. Nutr Cancer. 1996;26(3):365-80. doi: 10.1080/01635589609514492. PMID 8910918
- [Result] Rafter J. The effects of probiotics on colon cancer development. Nutr Res Rev. 2004 Dec;17(2):277-84. doi: 10.1079/NRR200484. PMID 19079931
- [Result] Saavedra JM, Bauman NA, Oung I, Perman JA, Yolken RH. Feeding of Bifidobacterium bifidum and Streptococcus thermophilus to infants in hospital for prevention of diarrhoea and shedding of rotavirus. Lancet. 1994 Oct 15;344(8929):1046-9. doi: 10.1016/s0140-6736(94)91708-6. PMID 7934445
- [Result] Sekine K, Toida T, Saito M, Kuboyama M, Kawashima T, Hashimoto Y. A new morphologically characterized cell wall preparation (whole peptidoglycan) from Bifidobacterium infantis with a higher efficacy on the regression of an established tumor in mice. Cancer Res. 1985 Mar;45(3):1300-7. PMID 3971375
- [Result] Sheng Y, Yang X, Lian Y, Zhang B, He X, Xu W, Huang K. Characterization of a cadmium resistance Lactococcus lactis subsp. lactis strain by antioxidant assays and proteome profiles methods. Environ Toxicol Pharmacol. 2016 Sep;46:286-291. doi: 10.1016/j.etap.2016.08.008. Epub 2016 Aug 6. PMID 27522548
- [Result] Smith PM, Howitt MR, Panikov N, Michaud M, Gallini CA, Bohlooly-Y M, Glickman JN, Garrett WS. The microbial metabolites, short-chain fatty acids, regulate colonic Treg cell homeostasis. Science. 2013 Aug 2;341(6145):569-73. doi: 10.1126/science.1241165. Epub 2013 Jul 4. PMID 23828891
- [Result] Stecher B. The Roles of Inflammation, Nutrient Availability and the Commensal Microbiota in Enteric Pathogen Infection. Microbiol Spectr. 2015 Jun;3(3). doi: 10.1128/microbiolspec.MBP-0008-2014. PMID 26185088
- [Result] Sun Y, O'Riordan MX. Regulation of bacterial pathogenesis by intestinal short-chain Fatty acids. Adv Appl Microbiol. 2013;85:93-118. doi: 10.1016/B978-0-12-407672-3.00003-4. PMID 23942149
- [Result] Tomkovich S, Jobin C. Microbiota and host immune responses: a love-hate relationship. Immunology. 2016 Jan;147(1):1-10. doi: 10.1111/imm.12538. Epub 2015 Nov 2. PMID 26439191
- [Result] Tsai TY, Chu LH, Lee CL, Pan TM. Atherosclerosis-preventing activity of lactic acid bacteria-fermented milk-soymilk supplemented with Momordica charantia. J Agric Food Chem. 2009 Mar 11;57(5):2065-71. doi: 10.1021/jf802936c. PMID 19216552
- [Result] Tsai YT, Cheng PC, Fan CK, Pan TM. Time-dependent persistence of enhanced immune response by a potential probiotic strain Lactobacillus paracasei subsp. paracasei NTU 101. Int J Food Microbiol. 2008 Dec 10;128(2):219-25. doi: 10.1016/j.ijfoodmicro.2008.08.009. Epub 2008 Aug 26. PMID 18809220
- [Result] Tuson HH, Weibel DB. Bacteria-surface interactions. Soft Matter. 2013 May 14;9(18):4368-4380. doi: 10.1039/C3SM27705D. PMID 23930134
- [Result] Van de Water J, Keen CL, Gershwin ME. The influence of chronic yogurt consumption on immunity. J Nutr. 1999 Jul;129(7 Suppl):1492S-5S. doi: 10.1093/jn/129.7.1492S. PMID 10395628
- [Result] Yu X, Li S, Yang D, Qiu L, Wu Y, Wang D, Shah NP, Xu F, Wei H. A novel strain of Lactobacillus mucosae isolated from a Gaotian villager improves in vitro and in vivo antioxidant as well as biological properties in D-galactose-induced aging mice. J Dairy Sci. 2016 Feb;99(2):903-914. doi: 10.3168/jds.2015-10265. Epub 2015 Dec 17. PMID 26709186